CLINICAL TRIAL: NCT06853067
Title: Effect of Dexmedetomidine and Remimazolam on Body Temperature in Patients Undergoing Spinal Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SMG-SNU Boramae Medical Center (Other)
Responsible Party: Principal Investigator, Jin-Young Hwang, MD., PhD, SMG-SNU Boramae Medical Center
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 20240701
Record Dates: First submitted 2025-02-18; First posted 2025-02-28 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Temperature Change, Body
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Dexmedetomidine is administered for sedation in patients undergoing spinal anesthesia
  Interventions: Other: Monitoring of body temperature
- Remimazolam group (Experimental): Remimazolam is administered for sedation in patients undergoing spinal anesthesia
  Interventions: Other: Monitoring of body temperature

INTERVENTIONS:
Other: Monitoring of body temperature — Body temperature is monitored in the forehead using the Temperature Monitoring Patient Sensors in patients sedated with dexmedetomidine or remimazolam during spinal anesthesia.

SUMMARY:
This study aims to evaluate the effect of dexmedetomidine and remimazolam on body temperature in patients undergoing spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for elective surgery under spinal anesthesia

Exclusion Criteria:

* Severe vascular disease
* Thyroid dysfunction
* Coagulopathy
* Neuromuscular disease.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2025-04-15 (Actual); Primary Completion 2025-08-28 (Actual); Study Completion 2025-08-28 (Actual)

PRIMARY OUTCOMES:
Incidence of hypothermia during surgery | Body temperature is monitored during surgery
  Incidence of temperature <36℃ during spinal anesthesia is assessed.

SECONDARY OUTCOMES:
Incidence of hypothermia in the post-anesthesia recovery room | Immediately after entering the the post-anesthesia recovery room, until the discharge
  Body temperature is assessed in the in the post-anesthesia recovery room
Incidence of shivering during surgery and in the post-anesthesia recovery room | During surgery and in the post-anesthesia recovery room
  Occurrence of shivering is assessed.

CONTACTS AND LOCATIONS:
Locations (1):
- SMG-SNU Boramae Medical Center, Seoul, Select State/Province, South Korea